CLINICAL TRIAL: NCT00861328
Title: A Phase 1 Dose-Escalation Study of the Safety and Clinical Effects of ON 01910.Na in Combination With Either Irinotecan or Oxaliplatin in Patients With Advanced Solid Tumors
Brief Title: Safety Study of ON 01910.Na in Combination With Irinotecan or Oxaliplatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-06
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Advanced Solid Tumors
Keywords: Phase 1; maximum tolerated dose; oxaliplatin; irinotecan; ON 01910.Na
MeSH Terms: interventions — ON 01910; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Treatment of escalating doses of ON 01910.Na in combination with irinotecan
  Interventions: Drug: ON 01910.Na and irinotecan
- B (Experimental): Treatment of escalating doses of ON 01910.Na in combination with oxaliplatin
  Interventions: Drug: ON 01910.Na and oxaliplatin

INTERVENTIONS:
Drug: ON 01910.Na and irinotecan — ON 01910.Na will be administered by IV infusion over 24 hours once per week in a 6-week cycle (6 doses per cycle). The dose of ON 01910.Na will start at 250 mg/m2 and will proceed to higher dose levels after safety evaluation.
  The suggested starting dose of Irinotecan is 180 mg/m2 administered by intravenous (IV) infusion over 90 minutes every 2 weeks of a 6-week cycle (3 doses per cycle). Reductions in the starting doses according to recommendations of current approved prescribing information may be considered after review of patients' medical histories and potential tolerances to treatment with the chemotherapy agent.
  Other Names: Campostar; camptothecin-11; irinotecan; irinotecan HCl; CPT-11; U-101440E; rigosertib sodium
  Arms: A
Drug: ON 01910.Na and oxaliplatin — ON 01910.Na will be administered by IV infusion over 24 hours once per week in a 6-week cycle (6 doses per cycle). The dose of ON 01910.Na will start at 250 mg/m2 and will proceed to higher dose levels after safety review of the combination regimen in the previous cohort.
  The suggested starting dose of Oxaliplatin is 85 mg/m2 administered by IV infusion over 120 minutes every 2 weeks of a 6-week cycle (3 doses per cycle). Reductions in the starting doses according to recommendations of current approved prescribing information may be considered after review of patients' medical histories and potential tolerances to treatment with the chemotherapy agent.
  Other Names: diaminocyclohexane oxalatoplatinum; oxalatoplatin; oxalatoplatinum; Eloxatin
  Arms: B

SUMMARY:
Treatment of cancer is often improved if two or more drugs are used in combination. In animal studies, the use of the combination of ON 01910.Na (a new, unapproved drug) and irinotecan or oxaliplatin (two approved and extensively used anti-cancer drugs) gave better results against tumor cells than the use of any of the single drugs alone. In addition, the use of the combinations did not result in an increase of side effects. This clinical trial will determine what is the highest dose of ON 01910.Na that can be given safely in combination with either irinotecan or oxaliplatin in human patients.

DETAILED DESCRIPTION:
This is an open-label, 2-arm, dose-escalation combination-therapy study in which patients with advanced malignancies will be assigned by the Investigator to dosing with either irinotecan plus ON 01910.Na (Group A), or oxaliplatin plus ON 01910.Na (Group B). The Investigator will make this assignment using clinical judgment, taking into consideration the patient's tumor type, UGT1A1 genotype when applicable (i.e., patients considered for treatment in Group A will be tested for UGT1A1 genotype, if not already known, and patients homozygous for the UGT1A1*28 allele will be excluded from Group A), prior treatment, and current clinical condition. Patients will be enrolled in 1 of 8 Cohorts (4 sequential Cohorts in Group A and 4 in Group B) of 3 patients each. Up to 6 additional patients will be tested at the MTD. Groups A and B will enroll and proceed simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years of age with histologically or cytologically confirmed solid tumors that are metastatic or progressive, for whom no standard therapy holds curative potential and for whom irinotecan or oxaliplatin are reasonable treatment options.
* Patients must have evaluable disease, either measurable on imaging or with informative tumor marker(s).
* Eastern Collaborative Oncology Group (ECOG) Performance Status of ≤2.
* Life expectancy >12 weeks.
* Any acute or chronic adverse effects of prior chemotherapy have resolved to <Grade 2 as determined by CTCAE v3 criteria.
* Existing or planned central venous access with a 2-channel infusion catheter system.
* Laboratory values meet the following criteria: Absolute neutrophil count ≥1,500 cells/µL; Platelets ≥100,000 cells/µL; Total bilirubin ≤1.5 times the upper limit of normal; AST (SGOT) ≤2.5 times the upper limit of normal; ALT (SGPT) ≤2.5 times the upper limit of normal; Serum creatinine ≤1.5 mg/dL or a measured creatinine clearance ≥50 mL/min; Negative βhCG test in women of childbearing potential (defined as women ≤50 years of age or history of amenorrhea for ≤12 months prior to study entry).
* Patients with primary liver cancer or hepatic metastasis are eligible to enroll, provided they meet the following: Total bilirubin is ≤2 mg/dL; AST and ALT are each ≤5 times the institutional upper limit of normal; Ascites, if present, is manageable with diuretic agents alone.
* If there is a history of treated brain metastases, these must have been clinically stable for ≥4 weeks prior to enrollment.
* UGT1A1 genotype of patient must be known or a UGT1A1 genotype test must be done for patients being considered for treatment in Group A.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Severe liver dysfunction (Child-Pugh Class C or uncompensated Class B with persistent encephalopathy, persistent ascites, or prothrombin time >1.5 times the upper limit of normal) is present.
* Patients with a history of esophageal bleeding are excluded unless varices have been sclerosed or banded and bleeding episodes have not occurred during the prior 6 months.
* Contraindications, including known hypersensitivity, to the assigned chemotherapy agent (i.e., irinotecan or oxaliplatin).
* Prior receipt of ON 01910.Na or prior participation in this protocol.
* Use of any investigational agents within 4 weeks of study enrollment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements, as determined by the Investigator.
* Patients who are homozygous for the UGT1A1*28 allele will be excluded from participating in Group A of this protocol.
* Patients with ascites requiring active medical management including paracentesis, peripheral bilateral edema or hyponatremia (defined as serum sodium value of <134 Meq/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 1 - 3 months

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 1 month
tumor measurements | 1 - 3 months
tumor markers | 1 - 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Mani, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Cancer Center, The Bronx, New York, United States

REFERENCES:
- [Background] Jimeno A, Chan A, Cusatis G, Zhang X, Wheelhouse J, Solomon A, Chan F, Zhao M, Cosenza SC, Ramana Reddy MV, Rudek MA, Kulesza P, Donehower RC, Reddy EP, Hidalgo M. Evaluation of the novel mitotic modulator ON 01910.Na in pancreatic cancer and preclinical development of an ex vivo predictive assay. Oncogene. 2009 Jan 29;28(4):610-8. doi: 10.1038/onc.2008.424. Epub 2008 Nov 24. PMID 19029951
- [Background] Jimeno A, Li J, Messersmith WA, Laheru D, Rudek MA, Maniar M, Hidalgo M, Baker SD, Donehower RC. Phase I study of ON 01910.Na, a novel modulator of the Polo-like kinase 1 pathway, in adult patients with solid tumors. J Clin Oncol. 2008 Dec 1;26(34):5504-10. doi: 10.1200/JCO.2008.17.9788. Epub 2008 Oct 27. PMID 18955447
- [Background] Reddy MV, Mallireddigari MR, Cosenza SC, Pallela VR, Iqbal NM, Robell KA, Kang AD, Reddy EP. Design, synthesis, and biological evaluation of (E)-styrylbenzylsulfones as novel anticancer agents. J Med Chem. 2008 Jan 10;51(1):86-100. doi: 10.1021/jm701077b. Epub 2007 Dec 19. PMID 18088089
- [Background] Gumireddy K, Reddy MV, Cosenza SC, Boominathan R, Baker SJ, Papathi N, Jiang J, Holland J, Reddy EP. ON01910, a non-ATP-competitive small molecule inhibitor of Plk1, is a potent anticancer agent. Cancer Cell. 2005 Mar;7(3):275-86. doi: 10.1016/j.ccr.2005.02.009. PMID 15766665
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- See also: Website of Albert Einstein Cancer Center. — http://www.aecom.yu.edu/cancer/